CLINICAL TRIAL: NCT05499780
Title: Post-market, Randomized and Controlled Clinical Study to Assess the Performance and Safety of Sentinox in the Prevention of Acute Respiratory Infections
Brief Title: Study on Performance and Safety of Sentinox in the Prevention of Acute Respiratory Infections (ARI)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrolment
Sponsor: APR Applied Pharma Research s.a. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STX-2022
Record Dates: First submitted 2022-08-08; First posted 2022-08-12 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: treatment with Sentinox performed 3 times/day for 21 days (Experimental): treatment with Investigational Medical Device (IMD) performed 3 times/day for 21 days at 8 am, 2 pm and 8 pm
  Interventions: Device: Sentinox
- Group B:no Sentinox treatment (No Intervention)

INTERVENTIONS:
Device: Sentinox — The treatment will be administered in a dose of 0.5 ml into each nostril (5 sprays) per 3 times/day (8 am, 2 pm and 8 pm), for 21 days from Visit 1.
  Arms: Group A: treatment with Sentinox performed 3 times/day for 21 days

SUMMARY:
This is a post market, single-center, randomized, controlled, clinical study to assessTo evaluate the performance of self-administered Sentinox intranasal spray in preventing ARI caused by at least one respiratory virus

DETAILED DESCRIPTION:
The study will consist of:

* A screening visit (Visit 0, on-site) to sign the informed consent form (ICF). The operator will:

  o review the inclusion/exclusion criteria

  o record the medical history, demographic data and concomitant medications (CMs), including previous anti-influenza, anti-COVID-19 and anti-pneumococcal vaccinations
* A randomization visit (Visit 1, on-site) to start the surveillance period. As soon as an increase in the regional epidemiological curve of ARI is observed, screened subjects will be invited for Visit 1. At Visit 1 the operator will:

  * check that the inclusion/exclusion criteria are still met, to confirm eligibility
  * confirm the medical history and the concomitant medications including previous anti-influenza, anti-COVID-19 and anti-pneumococcal vaccinations
  * record the result of the pregnancy testing
  * randomize with a 1:1 ratio in one of 2 trial Groups: - Group A: treatment with Investigational Medical Device (IMD) performed 3 times/day for 21 days at 8 am, 2 pm and 8 pm

    - Group B: no IMD treatment
  * invite the subjects to start: - treatment and surveillance period for 21 days, if belonging to Group A

    * surveillance period for 21 days, if belonging to Group B At Visit 1, an e-diary access will be delivered to both Groups to daily record Adverse Events (AEs), CMs other than treatments recorded in V1, presence of clinical features of ARI and IMD usage. The regular usage of the IMD will be recorded daily, as well as any change of the device and the reason for this. Study participants will install the Mobile App to complete the e-diary and will receive instructions to use the app. They will be instructed not to disclose their assignment to the treatment group to the blinded Investigator.

The IMD bottles needed for the 21-days treatment will be delivered to the enrolled participants of Group A, who will be trained to self-administer the treatment.

• A surveillance 21-days period, during which:

* the subjects of Group A will perform the daily treatment for 21 days
* the subjects of Group A and B will fill in a daily e-diary; the subjects will receive a reminder to follow the therapy (in the morning) and to complete the e-diary (in the evening)
* as soon as the subject records at least one symptom of ARI (i.e., cough, sore throat, shortness of breath, coryza as described in the European Commission guideline on relevant case definitions of communicable diseases [Commission Implementing Decision (EU) 2018/945 of 22 June 2018]) in the Mobile App, the blinded Investigator will be advised and will contact the subject by telephone within 12 hours to verify that the illness is due to ARI and to accordingly update the eCRF.

If during the phone contact the blinded Investigator judges the symptoms as correlated to ARI:

* the subject will be invited to immediately stop the IMD treatment if belonging to Group A
* the subject will be invited to the site for Visit 2 within 24 hours to perform a nasopharyngeal swab and to interrupt the surveillance period (Group A and B).

If during the phone contact the blinded Investigator judges the symptoms as not correlated to ARI, the subject will continue the surveillance period and the IMD treatment (if belonging to Group A) till a maximum of 21 days.

• A final visit (Visit 2, on-site). The subject, whose symptom of ARI during the surveillance period has been confirmed by the Investigator during the phone call, will attend for a site visit and be requested to:

* have a nasopharyngeal swab taken
* undergo a physical examination
* fill in the Visual Analogue Scale (VAS) score for Sentinox tolerability (for subjects of Group A)
* complete a 5-points Likert Scale for the satisfaction of Sentinox (for subjects of Group A)
* return the used and unused treatment bottles (for subjects of Group A)

The subject who does not have any symptom of ARI during the surveillance period, will perform a visit within 21±7 days from Visit 1 to:

* fill in the VAS score for Sentinox tolerability (for subjects of Group A)
* complete a 5-points Likert Scale for the satisfaction of Sentinox (for subjects of Group A)
* return the used and unused treatment bottles (for subjects of Group A) At Visit 2, the Mobile App will be uninstalled from the electronic device used by the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. ICF signed.
2. Males and females aged ≥ 18 years and <64 years at the time of the signature of the ICF.
3. Subjects who are willing to comply with the requirements of the study protocol, attend scheduled visits and calls for the duration of the study by telephone contact and install the Mobile App to use the e-diary.

Exclusion Criteria:

1. Reporting of any symptoms of ARI in the 15 days preceding the Visit 1.
2. Reporting the intake of any drugs, among antiviral or antibacterial therapies, that may interfere with the study results in the 15 days preceding the Visit 1.
3. Presence of any relevant organic, systemic or metabolic disease (particularly significant history of cardiac, renal, neurological, psychiatric, oncology, endocrinology, metabolic or hepatic disease).
4. Immune system illnesses.
5. Known drug and/or alcohol abuse.
6. Individuals who are cognitively impaired and/or who are unable to give informed consent.
7. Ongoing or prior participation in any other clinical trial of an experimental treatment within 30 days from Visit 1.
8. Concurrent or planned treatment with other agents with actual or possible direct antiviral/antibacterial activity.
9. Positive pregnancy test or breastfeeding woman.
10. Known hypersensitivity to the study treatment, its metabolites, or formulation excipient.
11. History of severe drug and / or food allergies.
12. Any condition that, in the opinion of the Investigator, would complicate or compromise the study or well-being of the Subject

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Performance of self-administered Sentinox intranasal spray in preventing ARI caused by at least one respiratory virus | Daily for a surveillance 21-days period
  Measure the proportion of patients with at least one symptoms of ARI (i.e., cough, sore throat, shortness of breath, coryza, as described in the European Commission guideline on relevant case definitions of communicable diseases [Commission Implementing Decision (EU) 2018/945 of 22 June 2018]) and confirmed by positive swab for at least 1 virus.

SECONDARY OUTCOMES:
Performance of Sentinox in preventing ARI caused by different respiratory viruses | Daily for a surveillance 21-days period
  Measure the Proportion of patients with at least one symptom of ARI (i.e., cough, sore throat, shortness of breath, coryza as described in the European Commission guideline on relevant case definitions of communicable diseases [Commission Implementing Decision (EU) 2018/945 of 22 June 2018]) and confirmed by positive swab for each specific strain of virus
Performance of Sentinox intranasal administration against bacterial infection | Daily for a surveillance 21-days period
  Measure the Proportion of patients with at least one symptom of ARI (i.e., cough, sore throat, shortness of breath, coryza as described in the European Commission guideline on relevant case definitions of communicable diseases [Commission Implementing Decision (EU) 2018/945 of 22 June 2018]), not confirmed by a positive swab for at least 1 virus, but with positive swab for at least 1 bacterium.
Performance of Sentinox in preventing clinically defined ARI without microbiological confirmation | Daily for a surveillance 21-days period
  Measure of Proportion of patients with at least one symptom of ARI (i.e., cough, sore throat, shortness of breath, coryza as described in the European Commission guideline on relevant case definitions of communicable diseases [Commission Implementing Decision (EU) 2018/945 of 22 June 2018]), not confirmed by positive swab for any of the tested virus or bacteria
Subjects' satisfaction of self -administering Sentinox | Daily for a surveillance 21-days period
  Measure the product satisfaction of subjects self-administering Sentinox by a 5-points Likert Scale
Tolerability and safety of Sentinox | Daily for a surveillance 21-days period
  Measure the Incidence and severity of AEs or incidents related to the use of the nasal solution, hypersensitivity and adverse reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Policlinico San Martino IRCCS, Genova, Italy